CLINICAL TRIAL: NCT02869750
Title: Evaluation of Adipokines ( Ghrelin, Resistin and Adiponectin), in Egyptian Women With Polycystic Ovary Syndrome
Brief Title: The Relationship Between Adipokines, Obesity and Insulin Resistance in Women With Polycystic Ovarian Syndrome
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, Lecturer in obstertics and gynecology, Ain Shams University Hospital, Ain Shams University
Other Study IDs: ADIPCOS
Record Dates: First submitted 2016-08-05; First posted 2016-08-17 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-02

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BLOOD SAMPLE
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obese PCOS: PCOS patients with BMI more than 25 kg/m2
- Lean PCOS: PCOS patients with BMI less than 25 kg/m2
- PCOS with normal HOMA2-1R: PCOS without Insuline resistance
- PCOS with elevated HOMA2-IR: PCOS with Insuline resistance

SUMMARY:
To evaluate possible clinical effects of adipokines , ( ghrelin, resistin and adiponectin), in obese and non-obese patients with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Seventy selected PCOS patients will be recruited for this study, and will be divided into two groups based on their body mass index (BMI): 35 obese (BMI≥ 25 kg/m2, group A), 35 non-obese (BMI<25 kg/m2, group B). In addition, 35 healthy non-obese women (BMI<25 kg/m2) will bw enrolled as the control (group C). Serum levels of FSH (follicle stimulating hormone), LH (luteinizing hormone), T(testosterone), glucose, insulin, adiponectin, resistin and resistin will bw detected, and compared the differences of them among three groups

ELIGIBILITY:
Inclusion Criteria:

* Females with PCOS in child bearing age who presented at reproductive and endocrinology clinics at Ain Shams University Maternity Hospital

Exclusion Criteria:

* Known androgen secreting tumor.
* PCO on ovarian stimulation medications
* PCO with any other medical illness.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females with PCOS in child bearing age who presented at reproductive and endocrinology clinics at Ain Shams University Maternity Hospital
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
serum ghrelin level | 24 hours
  measuring ghrelin, and ) in the three groups
serum resistin level | 24 hours
  serum resistin level in the three groups
serum adiponectin level | 24 hours
  serum adiponectin level in the three groups

SECONDARY OUTCOMES:
Glucose/Insulin ratio | 24 hours
  fasting glucose and insulin in three groups
serum testosterone level | 24 hours after labor
  serum testosterone level in three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Kotb, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided